CLINICAL TRIAL: NCT00833638
Title: Tadalafil 2.5 mg and 5 mg Once a Day Compared to Placebo in Day of Onset of Efficacy
Brief Title: A Study in Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12719; H6D-US-LVHZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tadalafil 2.5 mg (Experimental): No drug during baseline period, 2.5 mg for 14 days, then will continue at 5 mg for 14 days.
  Interventions: Drug: Tadalafil
- Tadalafil 5 mg (Experimental): No drug during baseline period, 5 mg for 14 days, then will continue at 5 mg for 14 days.
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): No drug during baseline period, placebo for 14 days, then will continue tadalafil at 5 mg for 14 days.
  Interventions: Drug: Placebo; Drug: Tadalafil

INTERVENTIONS:
Drug: Placebo — One tablet orally daily
  Arms: Placebo
Drug: Tadalafil — Orally once daily
  Other Names: Cialis; LY450190

SUMMARY:
The purpose of this study is to determine the day of onset of efficacy of tadalafil dosed once-a-day.

ELIGIBILITY:
Inclusion Criteria:

* Male and at least 18 years old, with at least a 3-month history of erectile dysfunction (ED).
* Anticipate having same adult female sexual partner during the study.
* Agree to make at least 4 sexual intercourse attempts with the female partner during the 4-week run-in phase without medication.
* Agree to make at least 1 sexual intercourse attempt per day with the female partner during days 1-4 following randomization (with a minimum of three attempts required during that period). Also agree to make at least 3 intercourse attempts during days 5-14 following randomization.
* Agree not to use any other ED treatment during the study and for 24 hours after the final study visit.

Partner Inclusion Criteria:

* Female and at least 18 years old.
* Agree to make at least 4 sexual intercourse attempts with the male sexual study partner during the 4-week run-in phase without medication.
* Agree to make at least 1 sexual intercourse attempt per day with the male partner during days 1-4 following randomization
* Agree to make at least 3 intercourse attempts during days 5-14 following randomization.

Exclusion Criteria:

* Previous or current treatment with tadalafil or any phosphodiesterase type 5 (PDE5) inhibitor on a daily basis for once daily use.
* ED caused by other primary sexual disorders, or untreated or inadequately treated endocrine disease.
* History of radical prostatectomy, other pelvic surgery or penile implant.
* Clinically significant penile deformity in the opinion of the investigator.
* Clinically significant renal insufficiency, or hepatobiliary disease as determined by the investigator.
* Glycosylated hemoglobin of >11%.
* Present with chronic stable angina treated with long-acting nitrates, or with chronic stable angina requiring short-acting nitrates in the last 90 days, or with angina occurring during sexual intercourse in the last 6 months.
* Have any significant cardiac conditions as described in the protocol exclusion criteria.
* Have a history of significant central nervous system injuries within the last 6 months.
* Have a history of Human Immunodeficiency Virus infection.
* Have any condition that would interfere with the subject's ability to provide informed consent or comply with study instructions, would place subject at increased risk, or might confound the interpretation of the study results.
* Currently receive treatment with nitrates, cancer chemotherapy, or antiandrogens (except finasteride taken as Propecia or Proscar, or Avodart [dutasteride]).
* History of drug, alcohol, or substance abuse within the past 6 months, as assessed by the investigator.
* Previously completed or withdrawn from any other study investigating tadalafil for once daily use.
* Received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Prior ineffective treatment with any PDE5 inhibitor in the opinion of the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first phase of the study was a run-in phase that lasted for approximately 4 weeks. During this time, subjects did not use any form of treatment for erectile dysfunction and were instructed to make at least 4 sexual intercourse attempts with their sexual partner. The purpose of this phase was to obtain baseline data for analysis purposes.
Period: Phase 2: Double-blind Treatment Phase
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Started | 121 | 118 | 133
Completed | 111 | 108 | 124
Not Completed | 10 | 10 | 9
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Entry Criteria Not Met | 3 | 2 | 1
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 3 | 3
Not completed — Sponsor Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2
Period: Phase 3: Open-label Extension Phase
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Started | 111 | 108 | 124
Completed | 110 | 105 | 122
Not Completed | 1 | 3 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo | Total
Number analyzed (Participants) | 121 | 118 | 133 | 372
Age Continuous [Mean (Standard Deviation); unit: years] | 59.63 (10.02) | 57.68 (11.07) | 59.23 (10.63) | 58.87 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 121 | 118 | 133 | 372
Race/Ethnicity, Customized [Number; unit: participants] — American Indian or Alaska Native
  participants
    American Indian or Alaska Native | 4 | 0 | 0 | 4
    Asian | 2 | 4 | 1 | 7
    Black or African American | 25 | 21 | 22 | 68
    Multiple | 1 | 6 | 2 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
    White | 89 | 87 | 107 | 283
Region of Enrollment [Number; unit: participants]
  United States | 121 | 118 | 133 | 372
Sexual Encounter Profile Diary question number 1 [Mean (Standard Deviation); unit: percentage of participants] — Sexual Encounter Profile Diary question number 1: "Were you able to achieve at least some erection (some enlargement of the penis)?" Data are presented as the mean percentage of participants who answered yes.
  percentage of participants | 74.04 (35.64) | 75.22 (35.69) | 82.26 (28.98) | 77.34 (33.55)
Sexual Encounter Profile Diary question number 2 [Mean (Standard Deviation); unit: percentage of participants] — Sexual Encounter Profile Diary question number 2: "Were you able insert your penis into your partner's vagina?" Data are presented as the mean percentage of participants who answered yes.
  percentage of participants | 52.70 (40.58) | 54.20 (39.47) | 56.16 (37.14) | 54.41 (38.94)
Sexual Encounter Profile Diary question number 3 [Mean (Standard Deviation); unit: percentage of participants] — Sexual Encounter Profile Diary question number 3: "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of participants who answered yes.
  percentage of participants | 30.90 (36.99) | 25.42 (32.62) | 29.95 (34.85) | 28.80 (34.85)
Sexual Encounter Profile Diary question number 4 [Mean (Standard Deviation); unit: percentage of participants] — Sexual Encounter Profile Diary question number 4: "Were you satisfied with the hardness of your erection?" Data are presented as the mean percentage of participants who answered yes.
  percentage of participants | 8.33 (19.18) | 4.96 (13.19) | 8.36 (16.88) | 7.26 (16.64)
Sexual Encounter Profile Diary question number 5 [Mean (Standard Deviation); unit: percentage of participants] — Sexual Encounter Profile Diary question number 5: "Were you satisfied overall with this sexual experience?" Data are presented as the mean percentage of participants who answered yes.
  percentage of participants | 7.67 (18.73) | 4.39 (12.31) | 8.08 (16.88) | 6.77 (16.27)

OUTCOME MEASURES:

1. Primary Outcome: Earliest Onset Day Measured by Cumulative Percentage of Participants With Yes Response to Sexual Encounter Profile Diary Question 3
Description: Cumulative percentage of participants achieving successful intercourse, as measured by "yes" responses to Sexual Encounter Profile diary question 3 (SEP3). SEP3 asks if the participant's erection lasted long enough to have successful intercourse.
Time Frame: 4 days during double-blind period
Population: Modified intent-to-treat population consisting of all participants who have at least 1 baseline observation and who took at least 1 dose of study drug followed by at least 1 intercourse attempt, and who recorded SEP diary data for it within the first 4 days of therapy following randomization.
Measure: Number; unit: cumulative percentage of participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 112 | 111 | 123
cumulative percentage of participants
  <= day 4 | 54.5 | 62.2 | 47.2
  <= day 3 | 49.1 | 55.0 | 42.3
  <= day 2 | 42.0 | 48.6 | 36.6
  <= day 1 | 28.6 | 25.2 | 28.5
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; The null-hypothesis was tested that there is no statistically significant difference in the onset of efficacy between tadalafil 2.5 mg and placebo as determined by the earliest day on which the cumulative percentage of subjects achieving at least 1 successful intercourse (within 4 days of starting treatment) is statistically significantly different between active drug and placebo; Test type: Superiority or Other; p = 0.086, Regression, Logistic — P-value for day <=4. A fixed-sequence test was used within each dose group at each time point (days 4, 3, 2, 1) and adjusted for multiple dose-placebo comparisons using the Bonferroni method. Testing started on day 4 and stopped when p>.025; Model response = treatment + pooled site + severity of erectile dysfunction at baseline
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; The null-hypothesis was tested that there is no statistically significant difference in the onset of efficacy between tadalafil 5 mg and placebo as determined by the earliest day on which the cumulative percentage of participants achieving at least 1 successful intercourse (within 4 days of starting treatment) is statistically significantly different between active drug and placebo; Test type: Superiority or Other; p = 0.006, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Model response = treatment + pooled site + severity of erectile dysfunction at baseline
Statistical Analysis 3: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.019, Regression, Logistic — P-value for day <=3. A fixed-sequence test was used within each dose group at each time point (days 4, 3, 2, 1) and adjusted for multiple dose-placebo comparisons using the Bonferroni method. Testing started on day 4 and stopped when p>.025; Model response = treatment + pooled site + severity of erectile dysfunction at baseline
Statistical Analysis 4: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.022, Regression, Logistic — P-value for day <=2. A fixed-sequence test was used within each dose group at each time point (days 4, 3, 2, 1) and adjusted for multiple dose-placebo comparisons using the Bonferroni method. Testing started on day 4 and stopped when p>.025; Model response = treatment + pooled site + severity of erectile dysfunction at baseline
Statistical Analysis 5: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.573, Regression, Logistic — P-value for day <=1. A fixed-sequence test was used within each dose group at each time point (days 4, 3, 2, 1) and adjusted for multiple dose-placebo comparisons using the Bonferroni method. Testing started on day 4 and stopped when p>.025

2. Secondary Outcome: Sexual Encounter Profile Diary Question Number 1, Change From Baseline to Post Baseline During the Double-blind Period in Percentage of Yes Responses
Description: Assessed was the mean change from baseline in the percentage of "yes" responses to the Sexual Encounter Profile Diary question number 1: "Were you able to achieve at least some erection (some enlargement of the penis)"? Data are presented as the mean percentage of participants who answered "yes".
Time Frame: Baseline and 14 days double-blind period
Population: Modified intent-to-treat population consisting of all subjects who have at least 1 baseline observation and who took at least 1 dose of study drug followed by at least 1 intercourse attempt, and who recorded SEP diary data for it within the first 4 days of therapy following randomization.
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 112 | 111 | 123
percentage of participants | 1.97 (2.33) | 2.74 (2.34) | -10.06 (2.24)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 1 exist between participants who received placebo and participants who received tadalafil 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; Included were terms for baseline value of the efficacy variable, treatment, site, and the baseline-by-treatment interaction were included; Mean Difference (Final Values) = 12.03, 95% CI 2-sided [5.72 to 18.34]
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 1 exist between participants who received placebo and participants who received tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; Terms for baseline value of the efficacy variable, treatment, site, and the baseline-by-treatment interaction were included; Mean Difference (Final Values) = 12.80, 95% CI 2-sided [6.48 to 19.12]

3. Secondary Outcome: Sexual Encounter Profile Diary Question Number 2, Change From Baseline to Post Baseline During the Double-blind Period in Percentage of Yes Responses
Description: Assessed was the mean change from baseline in the percentage of "yes" responses to the Sexual Encounter Profile Diary question number 2: "Were you able insert your penis into your partner's vagina?" Data are presented as the mean percentage of participants who answered yes.
Time Frame: Baseline and 14 days double-blind period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 112 | 111 | 123
percentage of participants | 8.11 (2.55) | 13.12 (2.56) | -7.29 (2.44)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 2 exist between participants who received placebo and participants who received tadalafil 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; Included were terms for baseline value of the efficacy variable, treatment, site, and the baseline-by-treatment interaction; Mean Difference (Final Values) = 15.40, 95% CI 2-sided [8.51 to 22.29]
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 2 exist between participants who received placebo and participants who received tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 20.41, 95% CI 2-sided [13.50 to 27.31]

4. Secondary Outcome: Sexual Encounter Profile Diary Question Number 3, Change From Baseline to Post Baseline During the Double-blind Period in Percentage of Yes Responses
Description: Assessed was the mean change from baseline in the percentage of "yes" responses to the Sexual Encounter Profile Diary question number 3: "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of participants who answered "yes".
Time Frame: Baseline and 14 days double-blind period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 112 | 111 | 123
percentage of participants | 15.67 (2.76) | 21.94 (2.77) | 1.40 (2.64)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 3 exist between participants who received placebo and participants who received tadalafil 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 14.27, 95% CI 2-sided [6.83 to 21.71]
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 3 exist between participants who received placebo and participants who received tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 20.54, 95% CI 2-sided [13.07 to 28.01]

5. Secondary Outcome: Sexual Encounter Profile Diary Question Number 4, Change From Baseline to Post Baseline During the Double-blind Period in Percentage of Yes Responses
Description: Assessed was the mean change from baseline in the percentage of "yes" responses to the Sexual Encounter Profile Diary question number 4: "Were you satisfied with the hardness of your erection?" Data are presented as the mean percentage of participants who answered "yes".
Time Frame: Baseline and 14 days double-blind period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 112 | 111 | 123
percentage of participants | 20.94 (2.90) | 28.50 (2.92) | 6.70 (2.77)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 4 exist between participants who received placebo and participants who received tadalafil 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 14.24, 95% CI 2-sided [6.42 to 22.06]
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 4 exist between participants who received placebo and participants who received tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 21.81, 95% CI 2-sided [13.94 to 29.67]

6. Secondary Outcome: Sexual Encounter Profile Diary Question Number 5, Change From Baseline to Post Baseline During the Double-blind Period in Percentage of Yes Responses
Description: Assessed was the mean change from baseline in the percentage of "yes" responses to the Sexual Encounter Profile Diary question number 5: "Were you satisfied overall with this sexual experience?" Data are presented as the mean percentage of participants who answered "yes".
Time Frame: Baseline and 14 days double-blind period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 112 | 111 | 123
percentage of participants | 20.45 (2.82) | 25.60 (2.84) | 6.52 (2.71)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 5 exist between participants who received placebo and participants who received tadalafil 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 13.92, 95% CI 2-sided [6.30 to 21.55]
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Tested was the null-hypothesis that no differences in the percentages of participants who answered "yes" to the sexual encounter profile diary question number 5 exist between participants who received placebo and participants who received tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiplicity; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 19.07, 95% CI 2-sided [11.40 to 26.75]

7. Secondary Outcome: Sexual Encounter Profile Diary Question 3, the Overall Distribution of Time to Onset by Yes Responses
Description: Assessed was the median time to onset of efficacy (day when 50% of participants have had at least 1 successful intercourse attempt) within the first 4 days of therapy based on a "yes" response to the sexual encounter profile diary question 3: "Did your erection last long enough for you to have successful intercourse?" Data are based on participants who responded "yes". For the placebo group, onset of efficacy was not reached within the first 4 days of therapy, therefore, the analysis timeframe was expanded for this group to determine the median time to onset of efficacy.
Time Frame: 4 days double-blind period
Population: Included in the analysis were all subjects with successful intercourse within the first 4 days of treatment, who have at least 1 baseline observation and who took at least 1 dose of study drug followed by at least 1 intercourse attempt, and who recorded SEP diary data for it within the first 4 days of therapy following randomization.
Measure: Median (Standard Error); unit: days
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 61 | 69 | 58
days | 4.0 (0.878) | 3.0 (0.384) | 6.0 (2.283)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Tested was the null-hypothesis that no differences in the time to onset of efficacy exists between participants who received placebo and participants who received tadalafil 2.5 mg, measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p = 0.301, Log Rank — No adjustment for multiplicity
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Tested was the null-hypothesis that no differences in the time to onset of efficacy exists between participants who received placebo and participants who received tadalafil 5 mg, measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p = 0.046, Log Rank — No adjustment for multiplicity

8. Secondary Outcome: Sexual Encounter Profile Diary Question 3, Daily Cumulative Percentage of Successful Intercourse Attempts
Description: Assessed was the cumulative precentage of successful intercourse attempts (successful attempts relative to the total number of intercourse attempts) over the 14-day double-blind treatment period. A successful attempt was defined by a "yes" response to the sexual encounter profile diary question #3: "Did your erection last long enough for you to have successful intercourse?" Data are presented as the proportion of intercourse attempts for which participants answered "yes" relative to the total number of intercourse attempts. Total number of attempts = TNA.
Time Frame: 14 days during double-blind period
Population: as for outcome 2
Measure: Number; unit: percentage of total number of attempts
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 112 | 111 | 123
percentage of total number of attempts
  <=day14 (TNA: n=905; n=813; n=781) | 45.1 | 46.6 | 30.9
  <=day13 (TNA: n=877; n=777; n=755) | 44.5 | 46.2 | 31.2
  <=day12 (TNA: n=827; n=730; n=711) | 44.0 | 45.9 | 30.8
  <=day11 (TNA: n=774; n=678; n=668) | 43.2 | 44.9 | 30.7
  <=day10 (TNA: n=726; n=626; n=625) | 41.9 | 44.2 | 30.6
  <=day9 (TNA: n=668; n=574; n=572) | 40.2 | 43.7 | 29.8
  <=day8 (TNA: n=608; n=534; n=523) | 39.5 | 42.8 | 29.6
  <=day7 (TNA: n=563; n=483; n=481) | 38.7 | 42.4 | 28.8
  <=day6 (TNA: n=505; n=439; n=435) | 37.4 | 41.6 | 27.9
  <=day5 (TNA: n=464; n=402; n=396) | 36.6 | 41.4 | 27.4
  <=day4 (TNA: n=412; n=350; n=352) | 37.1 | 40.9 | 26.2
  <=day3 (TNA: n=324; n=265; n=262) | 35.5 | 38.5 | 27.2
  <=day2 (TNA: n=214; n=179; n=175) | 35.8 | 38.9 | 28.0
  <=day1 (TNA: n=109; n=83; n=83) | 38.6 | 33.7 | 32.1
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Tested was the null-hypothesis that no differences in the precentage of successful intercourse attempts exists between participants who received placebo and participants who received tadalafil 2.5 mg, measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=14. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 2: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=13. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 3: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=12. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 4: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=11. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 5: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=10. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 6: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=9. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 7: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — P-value for day <=8. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 8: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.001, Regression, Logistic — P-value for day <=7. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 9: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — P-value for day <=6. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 10: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — P-value for day <=5. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 11: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — P-value for day <=4. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 12: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.009, Regression, Logistic — P-value for day <=3. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 13: Comparison: Tadalafil 2.5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.038, Regression, Logistic — P-value for day <=2. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 14: Comparison: Tadalafil 5 mg vs Placebo; Tested was the null-hypothesis that no differences in the proportion of successful intercourse attempts exists between participants who received placebo and participants who received tadalafil 5 mg, measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=14. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 15: Comparison: Tadalafil 5 mg vs Placebo; Tested was the null-hypothesis that no differences in the precentage of successful intercourse attempts exists between participants who received placebo and participants who received tadalafil 5 mg, measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=13. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 16: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=12. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 17: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=11. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 18: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=10. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 19: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=9. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 20: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=8. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 21: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=7. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 22: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=6. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 23: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=5. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 24: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for day <=4. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 25: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p = 0.003, Regression, Logistic — P-value for day <=3. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 26: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p = 0.008, Regression, Logistic — P-value for day <=2. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline
Statistical Analysis 27: Comparison: Tadalafil 5 mg vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p = 0.246, Regression, Logistic — P-value for day <=1. No adjustment for multiplicity; Response = Treatment + Pooled Site + Severity of ED at Baseline

9. Secondary Outcome: Sexual Encounter Profile Diary Question 3, Percentages of Yes Responses During the Double-blind and Open-label Periods for Participants Who Were Assigned to Placebo in the Double-blind Treatment Period
Description: Assessed were percentages of successful intercourse attempts relative to the total number of intercourse attempts over the 14-day open-label treatment period compared with the 14-day double-blind treatment period by dose group during the double-blind treatment period. A successful attempt was defined by a "yes" response to the sexual encounter profile diary question #3: "Did your erection last long enough for you to have successful intercourse?"
Time Frame: 14 days double-blind and 14 days open-label
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage successful attempts
Groups:
- Placebo Double-blind: No drug during baseline period, placeob for 14 days, then will continue at 5 mg for 14 days.
- Tadalafil 5 mg Open-label: No drug during baseline period, 5 mg for 14 days, then will continue at 5 mg for 14 days.
Arm/Group | Placebo Double-blind | Tadalafil 5 mg Open-label
Number analyzed (Participants) | 112 | 112
percentage successful attempts | 32.21 (35.35) | 68.27 (38.76)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Tadalafil 5 mg Open-label; Tested was the null-hypothesis that no differences in the proportion of successful intercourse attempts exist in patients who received placebo in the double-blind treatment period when comparing their proportion of succesful intercourse attempts between the double-blind treatment period (while receiving placebo) and the open-label treatment period (while receiving tadalafil 5 mg), measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -36.05 — the estimated mean difference shows changes in the double-blind treatment phase minus changes in the open label treatment phase

10. Secondary Outcome: Sexual Encounter Profile Diary Question 3, Percentages of Yes Responses in the Double-blind Period and the Open-label Period for Participants Who Were Assigned to Tadalafil 2.5 mg in the Double-blind Treatment Period
Description: as for outcome 9
Time Frame: 14-day double-blind and 14-day open-label
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage successful attempts
Groups:
- Tadalafil 2.5 mg Double-blind: No drug during baseline period, 2.5 mg for 14 days, then will continue at 5 mg for 14 days.
Arm/Group | Tadalafil 2.5 mg Double-blind | Tadalafil 5 mg Open-label
Number analyzed (Participants) | 101 | 101
percentage successful attempts | 46.11 (37.17) | 68.33 (40.10)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg Double-blind vs Tadalafil 5 mg Open-label; Tested was the null-hypothesis that no differences in the proportion of successful intercourse attempts exist in patients who received tadalafil 2.5 mg in the double-blind treatment period when comparing their proportion of succesful intercourse attempts between the double-blind treatment period (while receiving tadalafil 2.5 mg) and the open-label treatment period (while receiving tadalafil 5 mg), measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -22.22 — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Sexual Encounter Profile Diary Question 3, Percentages of Yes Responses in the Double-blind Period and the Open-label Period for Participants Who Were Assigned to Tadalafil 5 mg in the Double-blind Treatment Period
Description: as for outcome 9
Time Frame: 14-day double-blind and 14-day open-label
Population: Modified intent-to-treat population consisting of all subjects who have at least 1 baseline observation, who took tadalafil 5 mg during the double-blind treatment period, and who took at least 1 dose of tadalafil 5 mg followed by at least 1 intercourse attempt during the open-label period.
Measure: Mean (Standard Deviation); unit: percentage successful attempts
Groups:
- Tadalafil 5 mg Double-blind; Tadalafil 5 mg Open-label: No drug during baseline period, 5 mg for 14 days, then will continue at 5 mg for 14 days.
Arm/Group | Tadalafil 5 mg Double-blind | Tadalafil 5 mg Open-label
Number analyzed (Participants) | 99 | 99
percentage successful attempts | 49.54 (38.60) | 67.70 (38.98)
Statistical Analysis 1: Comparison: Tadalafil 5 mg Double-blind vs Tadalafil 5 mg Open-label; Tested was the null-hypothesis that no differences in the proportion of successful intercourse attempts exist in patients who received tadalfil 5 mg in the double-blind treatment period when comparing their proportion of succesful intercourse attempts between the double-blind treatment period (while receiving tadalafil 5 mg) and the open-label treatment period (while receiving tadalafil 5 mg), measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -18.16 — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Sexual Encounter Profile Diary Question 3, Percentages of Yes Responses During the Double-blind Period and the Open-label Period for Participants Who Didn't Respond to Tadalafil 2.5 mg During Double-blind Period
Description: Assessed were percentages of successful intercourse attempts relative to the total number of intercourse attempts in both treatment periods. A successful attempt was defined by a "yes" response to the sexual encounter profile diary question #3: "Did your erection last long enough for you to have successful intercourse?"
Time Frame: 14 days double-blind and 14 days open-label
Population: Modified intent-to-treat population consisting of all subjects who received tadalafil 2.5 mg in the double-blind study period and did not respond to treatment in that treatment period, who have at least 1 baseline observation and who took at least 1 dose of tadalafil 5 mg in the open-label period followed by at least 1 intercourse attempt.
Measure: Mean (Standard Deviation); unit: percentage successful attempts
Groups:
- Tadalafil 5 mg Open-label: No drug during baseline period, 2.5 mg for 14 days, then will continue at 5 mg for 14 days.
Arm/Group | Tadalafil 2.5 mg Double-blind | Tadalafil 5 mg Open-label
Number analyzed (Participants) | 49 | 49
percentage successful attempts | 32.51 (40.77) | 57.62 (45.27)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg Double-blind vs Tadalafil 5 mg Open-label; Tested was the null-hypothesis that no differences in the percentages of successful intercourse attempts exist in participants who received tadalafil 2.5 mg in the double-blind treatment period and did not respond to treatment when comparing their percentage of succesful intercourse attempts between the double-blind treatment period and the open-label treatment period (while receiving tadalafil 5 mg), measured by a response of "yes" to the sexual encounter profile diary question number 3; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -25.11 — [estimate comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Groups:
- Tadalafil 2.5 mg: No drug during baseline period followed by tadalafil 2.5 mg for 14 days.
- Tadalafil 5 mg: No drug during baseline period followed by tadalafil 5 mg for 14 days.
- Placebo: No drug during baseline period followed by placebo for 14 days.
- Tadalafil 2.5 mg to Tadalafil 5 mg: Participants receiving tadalafil 5 mg in the open-label period after receiving tadalafil 2.5 mg in the double-blind period.
- Tadalafil 5 mg to Tadalafil 5 mg: Participants receiving open-label tadalafil 5 mg after receiving tadalafil 5 mg in the double-blind period.
- Placebo to Tadalafil 5 mg: Participants receiving open-label tadalafil 5 mg after receiving placebo in the double-blind period.
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo | Tadalafil 2.5 mg to Tadalafil 5 mg | Tadalafil 5 mg to Tadalafil 5 mg | Placebo to Tadalafil 5 mg
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/118 | 0/133 | 0/111 | 0/108 | 0/124
Other Adverse Events (participants affected / at risk) | 13/121 | 12/118 | 8/133 | 6/111 | 9/108 | 4/124
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 2.5 mg (N=121) | Tadalafil 5 mg (N=118) | Placebo (N=133) | Tadalafil 2.5 mg to Tadalafil 5 mg (N=111) | Tadalafil 5 mg to Tadalafil 5 mg (N=108) | Placebo to Tadalafil 5 mg (N=124)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days